CLINICAL TRIAL: NCT05685901
Title: Ensayo clínico Aleatorizado y Controlado Para la evaluación de la Eficacia y Seguridad de la Inmunoprofilaxis orofaríngea Con Aceite de Oliva Rico en Polifenoles Como atenuación y prevención de la Enfermedad Infecciosa Por el Coronavirus SARS-CoV-2.
Brief Title: Oropharyngeal Immunoprophylaxis With High Polyphenolic Olive Oil as Clinical Spectrum Mitigating Factor in COVID-19.
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Nuestra Señora del Prado (Other)
Responsible Party: Principal Investigator, Francisco Rodríguez Argente, Head of Pediatric Department, Hospital General Nuestra Señora del Prado
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OLEOCOVID
Record Dates: First submitted 2023-01-10; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High polyphenolic olive oil (Experimental): Participants were required to take 2 mL of early harvest olive oil (normal early harvest olive oil) twice a day for three months and went through a clinical questionnaire at days 15, 30, 60 and 90. Participants were sent an envelope closed with instructions and informed consent. The primary outcome was to determine the effect of high polyphenolic olive oil on Coronavirus disease incidence, duration and severity. This study was approved by the independent ethic committee of the Hospital Nuestra Señora del Prado in Talavera de la Reina, belonging to the National Health System in Spain, and conducted in accordance with Declaration of Helsinki and Good Clinical Practice guidelines. Written informed consent was obtained from all patients. This questionnaire consisted in asking about having symptoms of SARS-CoV-2 infection, fever, low fever, malaise, headache, loss of smell, runny nose, sore throat.
  Interventions: Dietary Supplement: High polyphenolic olive oil. (Early harvest olive oil).
- No intervention (No Intervention): Participants were required to complete a questionnaire at days 15, 30, 60 and 90 of the study. This questionnaire consisted in asking about having symptoms of SARS-CoV-2 infection, fever, low fever, malaise, headache, loss of smell, runny nose, sore throat.

INTERVENTIONS:
Dietary Supplement: High polyphenolic olive oil. (Early harvest olive oil). — High polyphenolic olive oil is normal olive oil obtained from early harvest olives, this early harvest olive oil has been widely used for culinary purposes for centuries. The investigators wanted to study if oromucosal immunoprophylaxis with small quantities of high polyphenolic olive oil (2 mL of olive oil equivalent to 5 mg of polyphenols) adiministered twice a day could have clinical mitigating effects on the disease caused by SARS-CoV-2 infection.The primary outcome was to determine the effect of high polyphenolic olive oil on Coronavirus disease incidence, duration and severity.
  Arms: High polyphenolic olive oil

SUMMARY:
Immunomodulation of local immune response at the oropharyngeal mucosa can hypothetically activate mucosal immunity, which can difficult SARS-CoV-2 main immune evasion mechanisms in early stages of the disease and send an effective warning to the adaptive immune system. There are previous studies on immunotherapeutic management of upper respiratory tract infections with olive polyphenols. The investigators would like to study if participants following oromucosal immunomodulation with tiny quantities of high polyphenolic olive oil (early harvest olive oil) could have more possibilities to have less severe symptoms and a better outcome after SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and non-pregnant women were eligible if they had been in contact of recent COVID-19 diagnosed people and radomly allocated to olive oil group or not treatment at all group.

Exclusion Criteria:

1. Participation in other studies the 6 months before.
2. Pregnant women.
3. Inabilty to oral feeding.
4. Diagnosis of any pathology able to increase risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence. | 3 months.
  High polyphenolic olive oil immunoprophylaxis intervention and incidence of COVID-19.

SECONDARY OUTCOMES:
Duration- | 3 months
  Time to resolution of symptoms of COVID-19 in participants versus normal population.
Severity. | 3 months.
  Differences in severity of symptoms of COVID-19 between participants and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Rodríguez, Principal Investigator — Head of Pediatric Department.
Locations (1):
- Hospital Nuestra Señora del Prado, Talavera de la Reina, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Argente F, Alba-Dominguez M, Ortiz-Munoz E, Ortega-Gonzalez A. Oromucosal immunomodulation as clinical spectrum mitigating factor in SARS-CoV-2 infection. Scand J Immunol. 2021 Jan;93(1):e12972. doi: 10.1111/sji.12972. Epub 2020 Sep 18. PMID 32892403
- [Background] Greenberg SB. Update on rhinovirus and coronavirus infections. Semin Respir Crit Care Med. 2011 Aug;32(4):433-46. doi: 10.1055/s-0031-1283283. Epub 2011 Aug 19. PMID 21858748
- [Background] de Wit E, van Doremalen N, Falzarano D, Munster VJ. SARS and MERS: recent insights into emerging coronaviruses. Nat Rev Microbiol. 2016 Aug;14(8):523-34. doi: 10.1038/nrmicro.2016.81. Epub 2016 Jun 27. PMID 27344959
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Callow KA, Parry HF, Sergeant M, Tyrrell DA. The time course of the immune response to experimental coronavirus infection of man. Epidemiol Infect. 1990 Oct;105(2):435-46. doi: 10.1017/s0950268800048019. PMID 2170159
- [Background] Shi Y, Wang Y, Shao C, Huang J, Gan J, Huang X, Bucci E, Piacentini M, Ippolito G, Melino G. COVID-19 infection: the perspectives on immune responses. Cell Death Differ. 2020 May;27(5):1451-1454. doi: 10.1038/s41418-020-0530-3. Epub 2020 Mar 23. No abstract available. PMID 32205856
- [Background] Somerville V, Moore R, Braakhuis A. The Effect of Olive Leaf Extract on Upper Respiratory Illness in High School Athletes: A Randomised Control Trial. Nutrients. 2019 Feb 9;11(2):358. doi: 10.3390/nu11020358. PMID 30744092
- [Background] Brandtzaeg P. Secretory immunity with special reference to the oral cavity. J Oral Microbiol. 2013;5. doi: 10.3402/jom.v5i0.20401. Epub 2013 Mar 11. PMID 23487566
- [Background] Beilharz MW, Cummins MJ, Bennett AL, Cummins JM. Oromucosal Administration of Interferon to Humans. Pharmaceuticals (Basel). 2010 Jan 28;3(2):323-344. doi: 10.3390/ph3020323. PMID 27713254

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT05685901/Prot_SAP_ICF_000.pdf